CLINICAL TRIAL: NCT03341377
Title: An Observational Study for Establishing the Patient-reported Outcome-based Perioperative Symptom Management Cohort in Patients With Lung Cancer
Brief Title: Perioperative Symptom Study of Lung Cancer (CN-PRO-Lung 1)
Status: Completed | Type: Observational
Sponsor: Xiaojun Yang (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Sichuan Cancer Hospital and Research Institute (Other); Zigong No.1 Peoples Hospital (Other); Jiangyou People's Hospital (Unknown); Chengdu Third People's Hospital (Unknown); Chengdu Seventh People's Hospital (Unknown); Dazhu County People's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Xiaojun Yang, Clinical Professor and Principal Investigator, Sichuan Cancer Hospital and Research Institute
Organization: Sichuan Cancer Hospital and Research Institute (Other)
Other Study IDs: SCCHEC-02-2017-042
Record Dates: First submitted 2017-11-08; First posted 2017-11-14 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Patient-reported Outcomes
Keywords: utility parameter; patient-reported outcome; perioperative symptom management; lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung cancer surgical patients: Patient-reported symptom assessments in patients undergoing lung cancer surgery.

SUMMARY:
Investigators propose a multicenter prospective observational cohort study to develop and validate essential technical parameters for establishing the patient-reported outcome-based perioperative symptom management cohort in patients with lung cancer. With at least 300 patients with initial diagnosis of lung cancer and scheduled for surgery, this study will administer symptom assessments (MDASI-LC) and quality of life assessments (SIQOL) before surgery (typically within 3 days before surgery), daily after surgery (in hospital ≤ 14 days), and weekly after discharge, up to 4 weeks (±3 days) or the start day of postoperative oncologic treatment. In the upgraded research protocol, symptom and quality of life assessments (every 3 month for 1 year, every 6 month for 2-3 year, every 12 month for 4-5 year), as well as the follow-up of clinical outcomes will continue until 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Be pathologically or clinically diagnosed as primary lung cancer before surgery;
2. Plan to undergo a surgical procedure.

Exclusion Criteria:

1. Aged younger than 18;
2. Diagnosis of cognitive impairment or unable to understand the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients planning to undergo surgery
Sampling Method: Non-Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Perioperative symptom burden (severity, freqency and impact on daily functioning) measured by MDASI-LC | less than 6 weeks
  We will use MD Anderson Symptom Inventory lung cancer module (MDASI-LC) to longitudinally assess the perioperative symptom burden for lung cancer patients. The symptom burden will be profiled as symptom severity, frequency of moderate to severe symptom and its interference with daily functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Yang, MD, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (6):
- China (6):
  - Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan
  - Chengdu Seventh People's Hospital, Chengdu, Sichuan
  - Chengdu Third People's Hospital, Chengdu, Sichuan
  - Dazhu County People's Hospital, Dazhou, Sichuan
  - Jiangyou People's Hospital, Jiangyou, Sichuan
  - Zigong First People's Hospital, Zigong, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liao J, Hu X, Wei X, Dai W, Yu H, Tian X, Wang Y, Qin Q, Xu N, Li Y, Li Q, Shi Q, Liu X. Sex-related differences in postoperative patient-reported outcomes among lung cancer patients: a multicenter cohort study. BMC Cancer. 2025 Apr 29;25(1):800. doi: 10.1186/s12885-025-14191-z. PMID 40301835
- [Derived] Wei X, Yu H, King-Kallimanis B, Liu Y, Huang L, Dai W, Yang D, Zhou X, Li Q, Shi Q. Long-Term Function Recovery Following Upper Versus Lower Lobectomy for Lung Cancer: A Multicenter Longitudinal Cohort Study. Thorac Cancer. 2025 Jan;16(1):e15505. doi: 10.1111/1759-7714.15505. Epub 2024 Dec 13. PMID 39670353
- [Derived] Dai W, Xie S, Zhang R, Wei X, Wu C, Zhang Y, Feng W, Liao X, Mu Y, Zhou H, Cheng X, Jiang Y, He J, Li Q, Yang X, Shi Q. Developing and validating utility parameters to establish patient-reported outcome-based perioperative symptom management in patients with lung cancer: a multicentre, prospective, observational cohort study protocol. BMJ Open. 2019 Oct 28;9(10):e030726. doi: 10.1136/bmjopen-2019-030726. PMID 31662377